CLINICAL TRIAL: NCT06839833
Title: A Prospective, Interventional Study to Assess the Clinical Performance of the APOL1 Genotyping Clinical Trial Assay in the Intended Use Population and Environment
Brief Title: APOL1 Genotyping CTA Clinical Performance Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Almac Diagnostic Services LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SP2024001
Record Dates: First submitted 2025-02-10; First posted 2025-02-21 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: APOL1-mediated Kidney Disease

STUDY DESIGN:
Intervention Model Description: The study will use the APOL1 Genotyping CTA to test deoxyribonucleic acid (DNA) extracted from blood specimens to identify individuals who are homozygous or compound heterozygous for apolipoprotein L1 (APOL1) high-risk genotypes (G1 and G2). The individuals who are identified as being homozygous or compound heterozygous for the APOL1 high-risk genotypes are candidates for enrolment onto an pharmaceutical company-sponsored, Phase 2b clinical trial which is investigating the safety and efficacy of a synthetic antisense oligonucleotide (ASO) for the treatment of APOL1-mediated kidney disease (AMKD). I.e. The APOL1 Genotyping CTA being used interventionally as it is determining eligibility onto a trial, however not used to determine stratification into clinical trial cohorts.
Masking Description: Almac Diagnostic Services receives de-identified specimens only for inclusion in the clinical performance study. The clinical trial protocol describes the blinding and un-blinding procedures for the clinical trial and this responsibility lies with the pharmaceutical clinical trial sponsor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- APOL1 Genotyping (Other): All study participants will submit a blood specimen for APOL1 Genotyping CTA screening. The APOL1 Genotyping CTA will identify individuals who are homozygous or compound heterozygous for apolipoprotein L1 (APOL1) high-risk genotypes (G1 and G2). The individuals who are identified as being homozygous or compound heterozygous for the APOL1 high-risk genotypes are candidates for enrolment onto an pharmaceutical company-sponsored, Phase 2b clinical trial which is investigating the safety and efficacy of a synthetic antisense oligonucleotide (ASO) for the treatment of APOL1-mediated kidney disease (AMKD).
  Interventions: Diagnostic Test: APOL1 Genotyping

INTERVENTIONS:
Diagnostic Test: APOL1 Genotyping — The APOL1 Genotyping CTA will identify individuals who are homozygous or compound heterozygous for apolipoprotein L1 (APOL1) high-risk genotypes (G1 and G2). The individuals who are identified as being homozygous or compound heterozygous for the APOL1 high-risk genotypes are candidates for enrolment onto an pharmaceutical company-sponsored, Phase 2b clinical trial which is investigating the safety and efficacy of a synthetic antisense oligonucleotide (ASO) for the treatment of APOL1-mediated kidney disease (AMKD).

SUMMARY:
Clinical Performance Study SP2024001, is a prospective, interventional study to assess the clinical performance of the APOL1 Genotyping Clinical Trial Assay (CTA) in the intended use population and environment. The study will use the APOL1 Genotyping CTA to test deoxyribonucleic acid (DNA) extracted from blood specimens to identify individuals who are homozygous or compound heterozygous for apolipoprotein L1 (APOL1) high-risk genotypes (G1 and G2).The individuals who are identified as being homozygous or compound heterozygous for the APOL1 high-risk genotypes are candidates for enrolment onto an pharmaceutical company-sponsored, Phase 2b clinical trial which is investigating the safety and efficacy of a synthetic antisense oligonucleotide (ASO) for the treatment of APOL1-mediated kidney disease (AMKD).

ELIGIBILITY:
Inclusion Criteria:

* Study participants must be identified as a potential candidate for the pharmaceutical company- sponsored clinical trial by their physician based on the clinical trial inclusion criteria.
* Study participant has agreed to and signed the clinical trial Informed Consent Form (inclusive of risks related to the APOL1 Genotyping CTA).
* The study participant's specimen must be distributed to the device test site accompanied by a complete Test Request Form signed by the appropriate clinical trial site personnel.
* All participant specimens must meet predetermined specifications (e.g., undamaged, appropriate volume, appropriate specimen type, appropriate disease indication) for acceptance for testing by the device test site in accordance with established procedures.

Exclusion Criteria:

* Study participants will be excluded as a potential candidate for the pharmaceutical company -sponsored clinical trial by their physician based on the clinical trial exclusion criteria as assessed at screening visit 1.
* The study participant has not agreed to and signed the (Clinical Trial) Informed Consent Form.
* The study participant's specimen is distributed to the device test site without a complete Test Request Form.
* The study participant's specimen did not meet predetermined specifications for acceptance for testing by the device test site in accordance with established procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of APOL1 genotype result within the study population (G1/G2/G0), for participants' specimens tested using the APOL1 Genotyping CTA | Through study completion, approximately 1 year
  To utilize the APOL1 Genotyping CTA as a screening test to identify participants homozygous or compound heterozygous for high risk APOL1 genotypes (G1/G2) for inclusion in a Ph 2b trial

SECONDARY OUTCOMES:
Percentage of specimens submitted for APOL1 Genotyping CTA testing which meet device turn-around time (TAT) | Through study completion, approximately 1 year
  To demonstrate with objective evidence how the APOL1 Genotyping CTA will be expected to perform in routine clinical practice
Percentage of specimens submitted for APOL1 Genotyping CTA testing which meet laboratory TAT | Through study completion, approximately 1 year
  To demonstrate with objective evidence how the APOL1 Genotyping CTA will be expected to perform in routine clinical practice
Percentage of specimens submitted for APOL1 Genotyping CTA testing for which the device 'test was not ordered accurately (TNOA) | Through study completion, approximately 1 year
  To demonstrate with objective evidence how the APOL1 Genotyping CTA will be expected to perform in routine clinical practice
Percentage 'Specimens Not Accepted (SNA)' by the clinical laboratory(ies) for APOL1 Genotyping CTA testing | Through study completion, approximately 1 year
  To demonstrate with objective evidence how the APOL1 Genotyping CTA will be expected to perform in routine clinical practice
Percentage of Quality Control Failures | Through study completion, approximately 1 year
  To demonstrate with objective evidence how the APOL1 Genotyping CTA will be expected to perform in routine clinical practice
Percentage of corrected reports | Through study completion, approximately 1 year
  To demonstrate with objective evidence how the APOL1 Genotyping CTA will be expected to perform in routine clinical practice
Percentage of updated reports | Through study completion, approximately 1 year
  To demonstrate with objective evidence how the APOL1 Genotyping CTA will be expected to perform in routine clinical practice
Percentage homozygous or compound heterozygous for APOL1 high risk genotypes within the study population | Through study completion, approximately 1 year
  To determine the expected homozygous/ compound heterozygous APOL1 high risk genotype prevalence

OTHER OUTCOMES:
AE/SAE/ADE/UADE/SADE incident rate | Through study completion, approximately 1 year
  Identification of AEs/ SAEs/ADE/UADE/SADE or complications associated with the APOL1 Genotyping CTA (participant and operator) inclusive of root cause identification (e.g., Device deficiency)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kennedy, MD PhD FRCP, Principal Investigator — Almac Diagnostic Services Ltd
Locations (1):
- Almac Diagnostic Services LLC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD, inclusive of the APOL1 Genotyping Clinical Trial Assay result
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Start date March 2025 End date March 2027
Access Criteria: The results of the APOL1 Genotyping CTA will be returned to the requesting clinical site (inclusive of clinical trial investigator) and the pharmaceutical clinical trial sponsor. The clinical trial investigator may return the result, if requested by the participant with appropriate genetic counselling. The device study will utilize remote electronic data capture systems to store and transfer data. Transfer of device data from Almac Diagnostic Services to the pharmaceutical clinical trial sponsor or other 3rd parties will be governed by agreed data transfer agreements and in line with local regulations.